CLINICAL TRIAL: NCT01158144
Title: A Phase II Study of Endostar, Paclitaxel/Carboplatin and Radiotherapy in Patients With Non-resectable Locally Advanced Non-small Cell Lung Cancer
Brief Title: Concurrent Endostar, Paclitaxel/Carboplatin and Radiotherapy for Locally Advanced Non-small Cell Lung (RT0902)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Shenglin Ma, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH03
Record Dates: First submitted 2010-05-13; First posted 2010-07-08 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Locally advanced; Radiotherapy; Concomitant Chemotherapy; Endostar
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — endostar protein; Endostatins; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endostar (Experimental): Patients with non-resectable non-small Cell Lung Cancer will receive thoracic radiation therapy 60-66 Gy over 30-33 fractions and concurrent with Endostar 7.5 mg/m2 over 3 hours d1-14, Paclitaxel 50 mg/m2 weekly over 1 hour, Carboplatin AUC = 2 mg/mL/min over 30 min weekly. Followed by Endostar 7.5 mg/m2 d1-14,Paclitaxel 175 mg/m2 d1 and Carboplatin AUC = 5 mg/mL/min d1 every 3 weeks for 2 cycles as consolidation treatment.
  Interventions: Drug: Endostar
- Conctrol (Active Comparator): Patients with non-resectable non-small Cell Lung Cancer will receive thoracic radiation therapy 60-66 Gy over 30-33 fractions and concurrent with Paclitaxel 50 mg/m2 weekly over 1 hour, Carboplatin AUC = 2 mg/mL/min over 30 min weekly. Followed by Paclitaxel 175 mg/m2 d1 and Carboplatin AUC = 5 mg/mL/min d1 every 3 weeks for 2 cycles as consolidation treatment.
  Interventions: Drug: Paclitaxel/Carboplatin

INTERVENTIONS:
Drug: Endostar — Patients with non-resectable non-small Cell Lung Cancer will receive thoracic radiation therapy 60-66 Gy over 30-33 fractions and concurrent with Endostar 7.5 mg/m2 over 3 hours d1-14, Paclitaxel 50 mg/m2 weekly over 1 hour, Carboplatin AUC = 2 mg/mL/min over 30 min weekly. Followed by Endostar 7.5 mg/m2 d1-14,Paclitaxel 175 mg/m2 d1 and Carboplatin AUC = 5 mg/mL/min d1 every 3 weeks for 2 cycles as consolidation treatment.
  Other Names: Recombinant Human Endostatin
  Arms: Endostar
Drug: Paclitaxel/Carboplatin — Patients with non-resectable non-small Cell Lung Cancer will receive thoracic radiation therapy 60-66 Gy over 30-33 fractions and concurrent with Paclitaxel 50 mg/m2 weekly over 1 hour, Carboplatin AUC = 2 mg/mL/min over 30 min weekly. Followed by Paclitaxel 175 mg/m2 d1 and Carboplatin AUC = 5 mg/mL/min d1 every 3 weeks for 2 cycles as consolidation treatment.
  Other Names: PC
  Arms: Conctrol

SUMMARY:
Concomitant chemoradiotherapy is the standard treatment of locally advanced, non-resectable, non-small cell lung cancer (NSCLC). However, the optimal chemotherapy regimen is still controversial. The purpose of this study was to evaluate the efficacy and toxicity of a concomitant treatment using Endostar (Recombinant Human Endostatin), Paclitaxel/Carboplatin and radiotherapy for LA-NSCLC, and also assess its impact on patient Quality of Life (QoL) and progression-free survival (PFS).

DETAILED DESCRIPTION:
Patients with non-resectable non-small Cell Lung Cancer will receive thoracic radiation therapy 60-66 Gy over 30-33 fractions and concurrent with Endostar 7.5 mg/m2 over 3 hours d1-14, Paclitaxel 50 mg/m2 weekly over 1 hour, Carboplatin AUC = 2 mg/mL/min over 30 min weekly. Followed by Endostar 7.5 mg/m2 d1-14,Paclitaxel 175 mg/m2 d1 and Carboplatin AUC = 5 mg/mL/min d1 every 3 weeks for 2 cycles as consolidation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small cell lung cancer (squamous cell carcinoma, adenocarcinoma, large cell carcinoma and etc)
* Presence of measurable disease by RECIST
* stage IIIA or IIIB, non-resectable
* ECOG performance status 0-1
* No prior chemotherapy, radiation therapy to chest, immunotherapy, or biologic therapy .Patients must sign an informed consent indicating that they are aware of the .investigational nature of the study in keeping with the policy of the hospital.

Exclusion Criteria:

* Carcinoid tumor, small cell carcinoma of lung
* Patients with any distant metastasis
* History of another malignancy except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
* Any other morbidity or situation with contraindication for radiotherapy (e.g. active infection, myocardial infarction preceding 6 months, symptomatic heart disease including unstable angina, congestive heart failure or uncontrolled arrhythmias, immunosuppressive treatment)
* Pregnant or lactating women, women who has not taken test of pregnancy (within 7 days before the first administration) and pregnant women
* Women and men of childbearing potential who have no willing of employing adequate contraception Tumor EGFR wild

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
tumor response rate | 1 month after treatment.
  Response was analyzed according to the RECIST system, based on CT scans.

SECONDARY OUTCOMES:
overall survival | baseline to date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Shenglin Ma, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Sun XJ, Deng QH, Yu XM, Ji YL, Zheng YD, Jiang H, Xu YP, Ma SL. A phase II study of Endostatin in combination with paclitaxel, carboplatin, and radiotherapy in patients with unresectable locally advanced non-small cell lung cancer. BMC Cancer. 2016 Apr 11;16:266. doi: 10.1186/s12885-016-2234-0. PMID 27067521